CLINICAL TRIAL: NCT02247544
Title: A Phase II Study on Trabectedin in Advanced Retroperitoneal Leiomyosarcoma and Well Differentiated/Dedifferentiated Liposarcoma
Brief Title: Efficacy Study on Trabectedin in Retroperitoneal Leiomyosarcoma and Well Differentiated/Dedifferentiated Liposarcoma
Acronym: TRAVELL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISG-STS-TRAB-2012; 2012-005428-14 (EudraCT Number)
Record Dates: First submitted 2014-09-05; First posted 2014-09-25 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Liposarcoma; Leiomyosarcoma
Keywords: STS, leiomyosarcoma, liposarcoma, trabectedin
MeSH Terms: conditions — Liposarcoma; Leiomyosarcoma; Ichthyosis, X-Linked | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trabectedin (Experimental): Trabectedin will be administered intravenously at a dose of 1.5 mg/m2 or 1.3 mg/m2 (at investigator's discretion, with a top-dose of 2.6 total mg per cycle) as a 24-hour infusion once every 3 weeks (cycle day 1).
  Since trabectedin has no cumulative toxicities, treatment can be continued until progressive disease, major toxicity, patient's intolerance or unwillingness to continue treatment or medical decision by the responsible physician. In the subgroup of patients amenable to surgery, treatment will be reasonably continued until the best dimensional response.
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Trabectedin administered at a dose of 1.5 mg/m2 - 1.3 mg/m2 (at investigator's discretion, with a top-dose of 2.6 total mg per cycle) as a 24-hour continuous infusion via a central venous access until progressive disease, major toxicity, patient's intolerance, unwillingness to continue treatment, or medical decision by the responsible physician
  Other Names: Yondelis

SUMMARY:
This is an Italian, multicentre, single arm, phase II study, with an intra-patient comparison end point. This study aims at confirming the activity of the drug trabectedin as second/further line treatment in retroperitoneal leiomyosarcoma and well differentiated/dedifferentiated liposarcoma expressed in terms of slowing down tumour growth.

Another objective is to investigate this peculiar benefit of trabectedin in typical retroperitoneal sarcomas may be exploited to help multidisciplinary clinical decision-making in the management of retroperitoneal sarcomas

DETAILED DESCRIPTION:
Retroperitoneal soft-tissue sarcomas (R-STSs) are rare neoplasms, accounting for 10% to 15% of Soft Tissue Sarcomas (STSs), which represent 1-3% of all cancers. They may show different histological types, but the predominant ones in the retroperitoneal region are: leiomyosarcoma, liposarcoma. The most commonly encountered in the retroperitoneum is the well differentiated/dedifferentiated liposarcoma.

First-line chemotherapy usually consists of doxorubicin and/or ifosfamide. These two drugs are the most active agents in adult STSs, with a dose-response relationship and response rates between 20% and 50%. However, the sarcoma community is currently doubtful as to the activity of ifosfamide in the subgroup of leiomyosarcomas.

Trabectedin has been found to be mainly active in leiomyosarcoma and liposarcoma and is approved by European Medicines Agency (EMA) as second-line chemotherapy for STSs. Although the response rate observed in pre-registration studies did not exceed 10%, trabectedin provided disease control, with progression arrest rates exceeding 50% and Progression Free Survival (PFS) rates exceeding 20% at 6 months.

Since so far no phase II studies tested the activity of trabectedin in retroperitoneal sarcomas, this is the specific aim of this study.

Target population: Patients with previously treated, histologically confirmed, retroperitoneal leiomyosarcoma and well differentiated/dedifferentiated liposarcoma. Patients may be either unamenable to surgery or amenable but in whom the addition of medical treatment is considered clinically advisable.

Translational studies will be performed, with the aim of characterising the tumour biological features associated with different response patterns to trabectedin. These assessments will be done in 15-20 patients who will undergo surgery after trabectedin, comparing tumour tissue specimens collected before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or locally relapsed and/or metastatic disease (in case of local disease, surgery may be technically feasible or not, but the clinical judgment must be that medical therapy is indicated)
* Pathology specimens available for centralized review
* Age ≥ 18 years
* European Eastern Cooperative Oncology Group Personal Status (ECOG PS) ≤ 2
* One or more previous systemic treatments employing anthracyclines and ifosfamide (unless one or both are clinically contraindicated)
* Measurable disease, as defined by Response Evaluation Criteria In Solid Tumors (RECIST)
* A minimum of 3 weeks since any previous medical therapy
* Recovery from toxic effects of prior therapies to National Cancer Institute Common Toxicity Criteria (NCI CTC) Grade 1 or lower
* Adequate haematological, renal and liver functions
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women
* Prior exposure to trabectedin
* Peripheral neuropathy, Grade 2 or higher
* History of other malignancies (except for basal cell carcinoma or cervical carcinoma in situ, adequately treated), unless in remission for 5 years or more and judged of negligible potential of relapse
* Known central nervous system (CNS) metastases
* Active viral hepatitis or chronic liver disease
* Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within one year before enrolment, uncontrolled arterial hypertension or arrhythmias
* Active major infection
* Other serious concomitant illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-03; Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Growth Modulation Rate | From date of randomization until progressive disease, assessed up to 48 months
  The primary end point of the study will be the proportion of responders to trabectedin, based on the ratio, in each single patient, between PFS under trabectedin (PFS) and time to progression after previous chemotherapy treatment (TTP1).

SECONDARY OUTCOMES:
Objective response (OR) in the overall sample | From date of randomization until progressive disease, assessed up to 48 months
Pathological tumour response in the two eligible histological types, in patients undergoing surgery after treatment | From date of randomization until the best tumour dimensional response, assessed up to 48 months
PFS and OR in the two eligible histological types | From date of randomization until progressive disease, assessed up to 48 months
PFS in patients who undergo surgery after, or during, medical therapy and those who do not | From date of randomization until progressive disease, assessed up to 48 months
Number of patients with grade>=3 adverse drug reactions, number of serious adverse events related to study drug and number of patients who will experience at least one serious adverse event | From date of randomization until progressive disease, assessed up to 48 months
Efficacy of trabectedin in reducing cancer related pain | From date of randomization until progressive disease, assessed up to 48 months
  All patients will be administered a standardized questionnaire evaluating cancer related pain and use of antalgic medication.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo G. Casali, MD, Principal Investigator — IRCCS Fondazione Istituto Nazionale per la cura dei tumori di Milano
Locations (21):
- Italy (21):
  - Istituto Tumori Giovanni Paolo II, Bari, BA
  - Azienda Ospedaliera Giovanni Paolo XXIII, Bergamo, BG
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna, BO
  - A.O. Spedali Civili, Brescia, BS
  - Ospedale Oncologico A. Businco, Cagliari, CA
  - Azienda Ospedaliera S Croce e Carle, Cuneo, CN
  - Azienda Ospedaliera Sant'Anna, Como, CO
  - IRST IRCCS Meldola, Meldola, FC
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Centro di Riferimento Oncologico di Aviano, Aviano, PD
  - Istituto Oncologico Veneto, Padua, PD
  - Azienda Ospedaliera Universitaria Santa Chiara, Pisa, PI
  - Ospedale Misericordia e Dolce, Prato, PO
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - Istituto per la Ricerca e la Cura del Cancro di Candiolo, Candiolo, TO
  - Ospedale Gradenigo, Torino, TO
  - Azienda Ospedaliera Santa Maria, Terni, TR
  - Istituto Nazionale Tumori - IRCCS - Fondazione Pascale, Napoli